CLINICAL TRIAL: NCT02868541
Title: Assessment of Pharyngeal Carriage of Microorganisms Responsible for Transmissible Acute Respiratory Infections in HAJJ Pilgrims
Acronym: EMIRATH
Status: Completed | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2013-29
Record Dates: First submitted 2016-08-11; First posted 2016-08-16 (Estimated); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Acute Respiratory Infection
Keywords: microorganisms; pilgrim; hajj

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Haaj pilgrim: Patient that are showing at the traveler hospital health center requiring the mandatory Meningococcal vaccine ACYW135
  Interventions: Other: Naso pharyngeal swab

INTERVENTIONS:
Other: Naso pharyngeal swab — Naso pharyngeal swab

SUMMARY:
The objective of this project is to study the prevalence of viruses and bacteria responsible for transmissible acute respiratory infections in the respiratory tract of pilgrims returning from the trip. The patients included, will be the consultant pilgrims to the traveler health center, and before leaving for Hajj. Based on the results obtained in previous studies, it is estimated that 200 pilgrims will be included each year, 600 in total (inclusion period of 3 years). Respiratory secretions are then collected by nasal swab and throat (swab) prior to departure for the hajj. In return, patients will be reconvened systematic consultation to record medical events potentially encountered during the trip, and it will again be performed the same nasal swabs and throat. It will then be performed on these samples' return from hajj "molecular detection (PCR and RT-PCR) of 35 viruses and bacteria respiratory tropism: influenza (3), RSV (2), metapneumovirus (1), Coronavirus (4), Parainfluenzavirus (4), enteroviruses (4), rhinovirus (1), adenovirus (6) bocavirus, polyomavirus (2), pneumococcus, Bordetella pertussis, Mycoplasma pneumoniae, Chlamydophila pneumoniae, Haemophilus influenzae, Neisseria meningitidis and Coxiella burnetii. Samples "return of hajj" positive should be cultured for the isolation of the strain. For patients positive return, it will be done further research of these 35 viruses and bacteria on samples "start of hajj," the same method described above. In addition to this systematic consultation, and if symptoms return, the pilgrims will be seen in consultation for a diagnosis evaluation and therapeutic management.

This study will shed light on the acquisition of microorganisms respiratory tropism during the stay and on the potential risks associated with the circulation of these pathogens after the trip.

ELIGIBILITY:
Inclusion Criteria:

* All travelers presenting during the study period in the service of international vaccination for mandatory meningococcal ACYW135 vaccination ,
* Affiliated to a social security insurance regime
* Male or Female
* Aged over 18 years
* Having signed informed consent form
* able to understand and answer the study questions

Exclusion Criteria

* Patients aged under 18
* Patient whose protocol compliance seems unlikely to investigator
* Participant in another clinical trial or in exclusion period of a previous clinical trial,
* Unable to understand the nature and objectives of the study,
* Refusing to sign the informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Travelers pilgrims over 18 years leaving for the Hajj pilgrimage and consulting at the international vaccination service of the Public Assistance of Marseille Hositals for the mandatory meningococcal ACYW135 vaccination.
Sampling Method: Probability Sample
Enrollment: 905 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2019-09-06 (Actual)

PRIMARY OUTCOMES:
The number of new viruses and/or bacteria identified and characterized by respiratory and pharyngeal carriage among pilgrims between the departure and the return of Hajj | up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: Undecided